CLINICAL TRIAL: NCT05112562
Title: Attentional Bias Modification Training for E-cigarette Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20.172
Record Dates: First submitted 2021-09-22; First posted 2021-11-09 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: E-cigarette Use; Tobacco Use Cessation
MeSH Terms: conditions — Vaping; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized attentional bias modification training (Experimental)
  Interventions: Behavioral: Computerized attentional bias modification training
- Placebo attention control training (Placebo Comparator)
  Interventions: Behavioral: Placebo attention control training

INTERVENTIONS:
Behavioral: Computerized attentional bias modification training — In intervention is designed to train participants to disengage attention from potent e-cigarette cues and is based on the well-established attention retraining paradigm for other psychopathologies.
  Arms: Computerized attentional bias modification training
Behavioral: Placebo attention control training — This control training is very similar to the intervention's overall task structure and stimuli. The only difference is that the this control program is designed to exert no systematic manipulation on the attention deployment pattern between the two stimulus categories, thereby yielding no significant impact on the level of attentional bas toward ENDS-related cues
  Arms: Placebo attention control training

SUMMARY:
Aims are to (1) evaluate attentional bias to e-cigarette cues between the intervention and control groups at post-intervention as compared to the pre-intervention; and (2) test the feasibility and efficacy of the intervention at post-intervention. To accomplish these aims, a theory-driven parallel, controlled 2-arm randomized clinical trial will be conducted with young adult e-cigarette users (approximately N = 50). Outcomes are attentional bias to e-cigarette cues and abstinence outcomes including nicotine dependence, and arousal/urges for e-cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 29 years
* Those who use ENDS exclusively, not combining with other tobacco, for 3 consecutive months
* Those who own a smartphone.

Exclusion criteria:

* Current medication or psychosocial treatment for ENDS dependence
* Serious alcohol-use problems (≥ 26 points on the Alcohol Use Disorders Identification Test)
* Ophthalmic conditions impeding eye-tracking
* Current psychiatric/psychosocial treatment for other mental health disorders in the DSM-5 (e.g., schizophrenia)
* Pregnancy.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Attentional bias to e-cigarette cues measured by cueing task | Pre-training
  Attentional bias measured by time in milliseconds between cue and response in cueing task
Attentional bias to e-cigarette cues measured by cueing task | 1-month follow up
  Attentional bias measured by time in milliseconds between cue and response in cueing task
Attentional bias to e-cigarette cues measured by cueing task | 2-months follow up
  Attentional bias measured by time in milliseconds between cue and response in cueing task
Attentional bias to e-cigarette cues measured by cueing task | 4-months follow up
  Attentional bias measured by time in milliseconds between cue and response in cueing task

SECONDARY OUTCOMES:
Subjective urges for e-cigarette use | Pre-training
  Subjective urges for ENDS use measured by E-cigarette Use Patterns questionnaire)
Nicotine dependence | Pre-training
  Nicotine dependence measured by Penn State E-Cigarette Dependence Index
Subjective urges for e-cigarette use | 1-momnth follow up
  Subjective urges for ENDS use measured by E-cigarette Use Patterns questionnaire)
Nicotine dependence | 1-month follow up
  Nicotine dependence measured by Penn State E-Cigarette Dependence Index
Subjective urges for e-cigarette use | 2-momnth follow up
  Subjective urges for ENDS use measured by E-cigarette Use Patterns questionnaire)
Nicotine dependence | 2-month follow up
  Nicotine dependence measured by Penn State E-Cigarette Dependence Index
Subjective urges for e-cigarette use | 4-momnth follow up
  Subjective urges for ENDS use measured by E-cigarette Use Patterns questionnaire)
Nicotine dependence | 4-month follow up
  Nicotine dependence measured by Penn State E-Cigarette Dependence Index

CONTACTS AND LOCATIONS:
Overall Officials: Seok Hyun Gwon, PhD, RN, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No